CLINICAL TRIAL: NCT01840358
Title: Evaluation of the Frequency of Hypoglycemia at Initiation of Insulin Pump Therapy in Children With Type 1 Diabetes
Brief Title: Hypoglycemia at Initiation of Pump Therapy in Children With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Patricia Olivier, Pediatric endocrinologist, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HSJ-3638
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Type 1 Diabetes
Keywords: Hypoglycemias; Insulin pump; Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients starting pump therapy (Other)
  Interventions: Other: Observation of hypoglycemias frequency 3 days before and after pump initiation

INTERVENTIONS:
Other: Observation of hypoglycemias frequency 3 days before and after pump initiation

SUMMARY:
The purpose of this study is to determine if patients have more hypoglycemic episodes the first 3 days following pump start compared to their usual number of hypoglycemias with our actual pump initiation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes with follow-up at the CHU Sainte-Justine
* Patient about to start insulin pump therapy at the CHU Sainte-Justine
* Last HbA1c between 7.2 and 9.7%
* Informed and signed consent

Exclusion Criteria:

* Type 1 diabetes diagnosed less than 1 year ago WITH total daily dose of insulin < 0.5U/kg/day
* Home of the patient at more than 50km of the CHU Sainte-Justine
* Refusal to consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of hypoglycemias | 6 days
  Frequency of hypoglycemias defined as blood sugars < 4.0mmol/l

SECONDARY OUTCOMES:
Frequency of hyperglycemias | 6 days
  Frequency of hyperglycemias defined as blood sugars > 17.0mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: patricia Olivier, Md, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Manousaki D, Deladoey J, Geoffroy L, Olivier P. Continuous Subcutaneous Insulin Infusion in Children: A Pilot Study Validating a Protocol to Avoid Hypoglycemia at Initiation. Front Endocrinol (Lausanne). 2017 Apr 24;8:84. doi: 10.3389/fendo.2017.00084. eCollection 2017. PMID 28484424